CLINICAL TRIAL: NCT06198049
Title: Effects of Pilates Training Versus Balance Proprioception Exercises on Lower Extremity Function in Children With Hearing Impairment
Brief Title: Effects of Pilates and Balance Proprioception Exercises on Hearing Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0735
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Hearing Impaired Children
Keywords: Hearing Impairment; Balance; Pilates
MeSH Terms: conditions — Hearing Loss | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: This will be Randomized Clinical Trial to see the effect of Pilates Training versus Balance Proprioception exercises on lower extremity function in children with hearing impairment
Who Masked: Participant
Masking Description: Participants will get a separate protocols and possible efforts will be put to mask the both groups about their treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Training (Experimental): Group A 17 participants will receive Pilates training General rehabilitation exercises. Balance and strengthening exercises. Stretching exercises will be performed.Each exercises will be performed with ten repetition for three sessions per week.
  Interventions: Other: Pilates Training
- Balance Proprioception Exercises (Experimental): Group B 17 participants will receive balance Proprioception exercises. The training program will consist of 14 basic exercises on and off the balance board, with variations on each exercise. The program will be included four prescribed exercises: (a) exercise without any material, (b) exercise with a ball only, (c) exercise with a balance board only, and (d) exercise with a ball and a balance board. Also for gait and dynamic balance activity training use of Cobblestones walking mat that affects postural control. Walking task on the Cobblestone walking mat included: walking backward, walking sideways, and walking under dim light conditions. Mat walking time per session increased from 6 to 12 min during the acclimation period of the first two sessions and progressed gradually but incrementally to a maximum of 20 min per session over the 12 ensuing sessions.
  Interventions: Other: Balance Proprioception Exercises

INTERVENTIONS:
Other: Pilates Training — This group will receive Pilates training General rehabilitation exercises. Balance and strengthening exercises. Stretching exercises will be performed.Each exercises will be performed with ten repetition for three sessions per week
  Arms: Pilates Training
Other: Balance Proprioception Exercises — This group will receive balance Proprioception exercises. The training program will consist of 14 basic exercises on and off the balance board, with variations on each exercise. Mat walking time per session increased from 6 to 12 min during the acclimation period of the first two sessions and progressed gradually but incrementally to a maximum of 20 min per session over the 12 ensuing sessions.
  Arms: Balance Proprioception Exercises

SUMMARY:
Static balance is the ability to hold the body in a specific position and posture, while dynamic balance is the ability to maintain balance while moving. Vision, somatosensation, vestibular, and hearing are integrated to achieve balance Ethical committee approval will be obtained. A written consent will be taken from all subjects in the language best understood by them, after fulfilling the inclusion criteria, Patients age 10-14 years will be recruited through Randomized Clinical trial in which convenient sampling technique will be used. Group A 17 participants will receive Pilates training and group B 17 participants will receive balance Proprioception exercises. Pediatric balance scale and Lower Extremity Functional scale will be used .The result after statistical analysis will either show both treatments equally effective or not. Data will be calculated before and after treatment with the help of outcome measure tools.

DETAILED DESCRIPTION:
Static balance is the ability to hold the body in a specific position and posture, while dynamic balance is the ability to maintain balance while moving. Vision, somatosensation, vestibular, and hearing are integrated to achieve balance. Various strategies are available in physiotherapy for addressing imbalance. Pilates and other balance proprioception exercises may be used as part of a treatment plan, albeit this may vary depending on the etiology of the imbalance. Patients age 10-14 years will be recruited through Randomized Clinical trial in which convenient sampling technique will be used. 34 Participants will be included in this study. Group A 17 participants will receive Pilates exercises, after the initial evaluations, the individuals in the Clinical Pilates training group will be informed about the definition, goals and benefits of clinical Pilates, will be familiarized with the exercises and how to use the five key elements of clinical Pilates (head-neck location - shoulder location - chest cage location - central focus [neutral position] - how they should preserve and maintain breathing) and group B 17 participants will receive balance Proprioception exercises on balance board with different exercises. Pediatric Balance Scale and Lower Extremity Functional scale will be used. The result after statistical analysis will either show both treatments equally effective or not. The results will be analyzed on SPSS.

ELIGIBILITY:
Inclusion Criteria

* Both Gender will be included.
* Age 10-14 years.
* No history of lower extremity injuries or neuromuscular problems during the last 6 months
* Child's physical fitness level to ensure they can safely participate in Pilates and balance proprioceptive exercises.
* Children having Cochlear implant

Exclusion Criteria

* Patients will be excluded from the study if they had significant cardiac, pulmonary, or metabolic comorbidity or had an active disease that required therapy modification during the study.
* If pain will be developed in skeletal muscles after training.
* The presence of a neurologic disease, decompensated organ failure, intra-articular steroid injection or surgery in any joint, active synovitis, active arthritis psychiatric disease, and inability to understand and follow the prescribed exercise

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale | Six weeks
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
Lower Extremity Functional Scale | Six weeks
  This consists of 20 questions about a person's capacity to carry out daily chores. Clinicians can use the LEFS to assess patients' initial function, ongoing progress, and outcome, as well as to set functional goals. The maximum score is 80 points, indicating very high function. The minimum possible score is 0 points, indicating very low functions

CONTACTS AND LOCATIONS:
Overall Officials: Iqra khan, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahafza MT, Wilson WJ, Brauer S, Timmer BHB, Hickson L. A Systematic Review of the Effect of Hearing Aids on Static and Dynamic Balance in Adults with Hearing Impairment. Trends Hear. 2022 Jan-Dec;26:23312165221121014. doi: 10.1177/23312165221121014. PMID 36377351